CLINICAL TRIAL: NCT02670759
Title: Continuous Thoracic Paravertebral Analgesia for Video-assisted Thoracoscopic Surgery (VATS): Analgesic Effectiveness and Role in Fast-track Surgery
Brief Title: Continuous Thoracic Paravertebral Analgesia for Video-assisted Thoracoscopic Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: A 30% decrease in opioid use was obeserved in the paravertebral analgesia group.
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15.291
Record Dates: First submitted 2016-01-18; First posted 2016-02-02 (Estimated); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paravertebral analgesia (Experimental): A paravertebral nerve block will be performed under ultrasound guidance by the anaesthesiologist prior to the induction of general anesthesia. A catheter will be inserted and a continuous infusion of bupivacaine will be administered.
  Interventions: Drug: Continuous infusion of bupivacaine
- Intercostal analgesia (Active Comparator): An intercostal nerve block using a single dose of bupivacaine will be performed by the surgeon at the end of surgery before skin closure.
  Interventions: Drug: Single dose of bupivacaine

INTERVENTIONS:
Drug: Continuous infusion of bupivacaine — The infusion of local anesthetics will be initiated using a conventional infusion pump and will be transferred on a portable elastomeric pump before discharge from the hospital if the patient is discharged the day after surgery or at the latest on the second morning following surgery. The infusion will continue on the portable pump for 30 hours.
  Arms: Paravertebral analgesia
Drug: Single dose of bupivacaine — A single dose of bupivacaine will be administered at the end of surgery before skin closure.
  Arms: Intercostal analgesia

SUMMARY:
This study is designed to assess:

* The impact of continuous thoracic paravertebral nerve blockade compared to intercostal nerve blockade on the intensity of postoperative pain following VATS in subjects having a Patient Controlled Analgesia (PCA) device as their primary analgesic modality.
* The impact of continuous thoracic paravertebral analgesia on length of stay, opioid intake, respiratory function, incidence of side-effects and postoperative complications.

The basic hypothesis of this study is that continuous thoracic paravertebral nerve blockade will provide superior postoperative analgesia following VATS when compared to intercostal nerve blockade in patients having a PCA device as their primary analgesic modality. Superior quality of analgesia should contribute to preserve pulmonary function, reduce opioid intake and related side-effects and shorten the hospital stay.

DETAILED DESCRIPTION:
Appropriate postoperative analgesia is crucial in fast-track surgery, which is a multimodal therapeutic strategy that aims toward enhanced postoperative recovery and shortened hospital stay. Although VATS is considered a minimally invasive procedure, patients have reported moderate to severe pain of variable duration following surgery. The ideal postoperative analgesia regimen for VATS has not been elucidated. Systemic opioids given through patient-controlled devices (PCA) are routinely used after these procedures but their analgesic effect can be limited and undesirable side-effects may occur. Intercostal nerve blockade is also widely used to alleviate pain following VATS and can be used as an adjunct to systemic opioids. Paravertebral nerve blockade is an interesting alternative for analgesia following VATS. The duration of pain relief associated with paravertebral nerve blockade may vary from 4 to 48 hours. However, the duration of the analgesic effect can be prolonged using a continuous infusion of local anesthetics.

This study will compare the efficacy of continuous ambulatory paravertebral analgesia to intercostal analgesia. All patients will have a PCA device as their primary analgesic modality.

Methods:

Seventy patients will be randomized to receive either continuous paravertebral analgesia or intercostal analgesia. Anesthetic technique and monitoring will be standardized.

On arrival in the recovery room, each patient will have a PCA device installed. PCA doses will be standardized. All patients will also receive acetaminophen and non-steroidal anti-inflammatory drugs (NSAIDS) as co-analgesia. PCA will be removed 24 hours after surgery and oral opioids will then be administered as needed.

From their arrival in the recovery room, patients in the paravertebral analgesia group will be administered a bupivacaine 0.0625% infusion through a conventional infusion pump at a rate of 10 mL/h. Before discharge from the hospital on the day following surgery or at the latest on the morning of the second day, the bupivacaine infusion will be transferred to a portable elastomeric pump. The infusion will continue for the next 30 hours at a rate of 10 mL/h.

During the first 72 hours following surgery, the following information will be recorded: intensity of pain, opioid intake, side-effects attributable to analgesia and patient's level of satisfaction towards pain management. The occurence of pulmonary complications will be noted. Lung function will be measured using a peak flow meter. Length of stay in the recovery room, in the intermediate intensive care unit and in the hospital will be recorded. Time to reach post-anesthesia discharge criteria will be recorded.

Patients will be contacted by telephone 2 times a day if hospital discharge occurs before 72 hours after surgery to assess their level of pain and analgesic intake, the presence of side-effects or complications and their satisfaction level towards pain management.

This trial will also include a sub-study to be performed on ten human cadavers. The goal of the sub-study will be to assess the impact of the orientation of the bevel of the paravertebral block needle on the ease of insertion and positioning of the paravertebral catheter using ultrasound imaging.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for an elective or emergency VATS surgery (lobectomy or bilobectomy)
* Patients eligible for fast-track surgery
* American Society of Anesthesiologists (ASA) physical status from 1 to 3

Exclusion Criteria:

* Contraindication to paravertebral nerve blockade
* Severe hepatic insufficiency
* Renal insufficiency
* Known allergy to local anesthetics, morphine or hydromorphone
* Contraindication to acetaminophen or non-steroidal anti-inflammatory drugs (NSAID)
* Inability to understand a verbal numeric pain scale despite previous instruction
* Inability to understand the instructions and precautions related to the use of a portable infusion pump or absence of a resource person or natural caregiver at home
* Preexisting pain at the site where the surgical incision will be made
* Current use of opioids, anticonvulsants or tricyclic antidepressants
* Recent history of drug or opioid abuse

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
Intensity of postoperative pain | 24 hours following surgery
  Will be assessed using a Verbal Numeric Pain Scale (VPNS) from 0 to 10: 0 being no pain at all and 10 being the worst pain imaginable

SECONDARY OUTCOMES:
Opioid intake | From surgery until 72 hours following surgery
Side-effects attributable to analgesia | From surgery until 72 hours following surgery
  The presence of nausea and vomiting will be recorded
Patient's satisfaction with pain relief | Daily from surgery until 72 hours following surgery
  Will be assessed using a scale from 1 to 4: 1 being completely dissatisfied and 4 being completely satisfied
Length of stay in the recovery room | At discharge from recovery room, approximately 1 hour after end of surgery
Length of stay in the intermediate intensive care unit | From discharge from the recovery room until discharge from the intermediate intensive care unit, approximately one day.
Length of stay in the hospital | From surgery until discharge from the hospital, approximately 2 days
Lung function | Immediately prior to surgery and daily from surgery until discharge from the hospital, approximately 2 days
  Will be measured using a peak flow meter
Pulmonary complications | From surgery until 72 hours following surgery
  Occurence of atelectasis or pneumonia will be noted
Time to reach discharge criteria | From the day after surgery until discharge from the hospital, approximately 2 days
  Will be assessed using the Post Anesthesia Discharge Score (PADS)
Intensity of postoperative pain | 48 hours following surgery
  Will be assessed using a Verbal Numeric Pain Scale (VPNS) from 0 to 10: 0 being no pain at all and 10 being the worst pain imaginable
Intensity of postoperative pain | 72 hours following surgery
  Will be assessed using a Verbal Numeric Pain Scale (VPNS) from 0 to 10: 0 being no pain at all and 10 being the worst pain imaginable

CONTACTS AND LOCATIONS:
Overall Officials: Sebastien Garneau, MD, FRCPC, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No